CLINICAL TRIAL: NCT04237545
Title: A Prospective, Randomized, Clinical Study of the Safety, Efficacy and Clinical Benefits of the T3® Short Dental Implant System Placed in the Posterior Regions
Brief Title: A Clinical Study of the T3 Short Dental Implant System
Acronym: Magnolia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1801
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous | interventions — Prostheses and Implants

STUDY DESIGN:
Intervention Model Description: The patient will be randomized to receive either the T3 short (test device) or the T3 standard length, ≥10mm, (control device) implant.
Who Masked: Investigator
Masking Description: The randomization will be done using assignment from a computerized algorithm program. This will be done using a fixed block randomization scheme to ensure 1:1 ratio between test and control groups. Sealed envelopes containing randomization cards (code) will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- T3 short implant (Experimental): The short implants are available in lengths of 5mm and 6mm and in diameters of 5mm and 6mm. For study both configurations, T3 short without nano-scale Discrete Crystalline Deposition (non DCD- surface treatment) and T3 short with nano-scale Discrete Crystalline Deposition (with DCD- surface treatment), will be used.
  Interventions: Device: T3 short and restoration (prosthesis)
- T3 standard length (Active Comparator): The T3 external hex implants available for this study will consist of lengths of 10mm, 11.5mm, 13mm, 15mm, 18mm and diameters of 4mm, 5mm, and 6mm. They have integrated platform switching (medialized implant/abutment junction). For study both configurations, T3 without nano-scale Discrete Crystalline Deposition (non DCD- surface treatment) and T3 with nano-scale Discrete Crystalline Deposition (with DCD- surface treatment), will be used.
  Interventions: Device: T3 standard length and restoration (prosthesis)

INTERVENTIONS:
Device: T3 short and restoration (prosthesis) — A qualified patient will be treated with a T3 short implant according to randomization assignment during implant placement surgery visit. The implant will then be restored with a prosthesis and followed up for yearly visits for a total of 4 years.
  Other Names: T3 short, T3
  Arms: T3 short implant
Device: T3 standard length and restoration (prosthesis) — A qualified patient will be treated with a T3 standard length implant according to randomization assignment during implant placement surgery visit. The implant will then be restored with a prosthesis and followed up for yearly visits for a total of 4 years.
  Other Names: T3
  Arms: T3 standard length

SUMMARY:
This clinical study will evaluate the safety and performance of the T3 short dental implant when placed in the posterior maxilla and mandible.

DETAILED DESCRIPTION:
This is a prospective, randomized-controlled, multicenter study in which patients in need of dental implants in the posterior maxilla and mandible will be treated with either the T3 short implant (test device) or the T3 standard length implant (control device). Qualified patients will have one or more edentulous areas in the posterior region to be restored using a single crown. All implants will be placed using a single-stage surgical protocol. A provisional or definitive (final) prosthesis will be placed (cemented or screw-retained) within 8 weeks of implant placement. All prosthetic work must be completed no later than 6 months following implant placement surgery.

Each site will be selected to place implants (both test and control) in either the DCD or the non-DCD configuration (a total of 30 implants per site). Among all study sites, a total of 120 implants (60 test, 60 control) will be enrolled in this study (any geographic region). The patient will be randomized to receive either the T3 short (test device) or the T3 standard length, ≥10mm, (control device) implant. Only patients meeting the inclusion / exclusion criteria and providing informed consent form will be enrolled into study. The duration of the study will be approximately 4 years from initiation to completion of data analysis and reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex and at least 18 years of age
2. Patients for whom a decision has already been made to use a dental implant for the restoration of existing partial edentulism in the posterior mandible or maxilla.
3. Prior extracted sites (at least 4 months after extraction) preferred; immediate extractions allowed
4. Splinting to a natural tooth is allowed for the short length (test) implants
5. Intact buccal table as verified by CBCT or during surgery. If absent, patient should be excluded from enrollment in the study.
6. Presence of opposing dentition (antagonist) that will allow for functional occlusion.
7. The site intended for implant placement should have a minimum amount of keratinized gingiva of 2mm and a sufficient vertical bone height (8 - 10 mm in the maxilla; 10mm in the mandible); a short implant (as determined by randomization) will be placed without the need for augmentation except for minor dehiscence, which can be augmented with autogenous bone chips to improve soft tissue attachment. If site was randomized to long length implant (control) (with a minimum of 8mm vertical bone height in the maxilla or less than 10 mm in the mandible) it will have simultaneous augmentation procedure (sinus elevation in the maxilla; vertical ridge augmentation in the mandible).
8. The site intended for implant placement should have approximately 1.5mm buccal-lingual distance on each side in order to allow for wide platform implant (5 and 6mm diameter).
9. Patients must be physically able to tolerate conventional surgical and restorative procedures.
10. Patients who provide a signed informed consent
11. Patients who agree to be evaluated for each study visit.

Exclusion Criteria:

1. Patients with known systemic diseases such as uncontrolled diabetes, endocrine disease, heart disease, immuno-compromised, or mental disorders.
2. Patients with current use of non-steroidal anti-inflammatory drugs, bisphosphonates or corticosteroid treatments.
3. Patients with active infection or severe inflammation in the areas intended for treatment.
4. Patients with a > 10 cigarette per day smoking habit.
5. Patients with a history of therapeutic radiation to the head or jaw.
6. Patients receiving other dental treatment(s) during the study that could have a negative impact on the healing phase of the study treatment sites.
7. Patients who are known to be pregnant at the screening visit or planning to become pregnant within 6 months of study enrollment.
8. Patients with evidence of severe parafunctional habits such as bruxing or clenching.
9. Patients who have previously failed dental implants at the site intended for study implant placement
10. Patients with HIV or Hepatitis infection
11. Patients with a history of generalized severe chronic periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Crestal Bone regression | 4 years
  Assess and compare peri-implant crestal bone level changes between test and control device from baseline to 4 years

SECONDARY OUTCOMES:
Implant integration and survival | 4 years
  Assess and compare integration success (mobility and ISQ assessments) between test and control device from baseline to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Hai Bo Wen, PhD, Study Director — ZimVie
Locations (4):
- United States (2):
  - Dr. Xiaozhe Han, Boston, Massachusetts
  - Dr. Suheil Boutros, Dearborn Heights, Michigan
- Dr. Stefano Sivolella, Padua, Italy
- Dr. Jordi Gargallo, Tarragona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No